CLINICAL TRIAL: NCT06153875
Title: Effects of Percutaneous Peripheral Nerve Stimulation on Neck and Low Back Pain: a Quadruple-blinded, Randomized Clinical Trial
Brief Title: Effects of Percutaneous Peripheral Nerve Stimulation on Neck and Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Francisco Ortega Rehabilitacion Avanzada SL (Other)
Collaborators: Ionclinics & DEIONICS. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPTE/2023-TBS
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Neck Pain; Low Back Pain
Keywords: Percutaneous peripheral nerve stimulation; Sensorimotor effects; Neck pain; Transcutaneous electrical nerve stimulation; Theta burst stimulation; Low back pain
MeSH Terms: conditions — Neck Pain; Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Randomised quadruple-blind clinical trial, with three intervention groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The order of the interventions will be randomized by a third person not involved in the treatment, assessment or statistical analysis. Once the care provider has inserted the needle in each subject, another third person will choose the protocol assigned on the stimulator, previously programmed and codified. Another investigator will take measurements of the variables of interest. Thus, nobody (participant, care provider, investigator and the outcome assessor) will know what intervention is applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sensory Threshold, Burst High Frequency (Experimental): The technique consists of percutaneous peripheral electrical stimulation on the Spinal or Inferior Gluteal and Tibial Nerve through a ultrasound-guided needle.
  Interventions: Other: Sensory Thresold, Burst High Frecuency
- Theta-Burst Stimulation (Experimental): The technique consists of percutaneous peripheral electrical stimulation on the Spinal or Inferior Gluteal and Tibial Nerve through a ultrasound-guided needle.
  Interventions: Other: Theta-Burst Stimulation
- Transcutaneous Electrical Nerve Stimulation (Active Comparator): The technique consists of transcutaneous electrical nerve stimulation on the trapezius or low back and internal calf muscles through surface electrodes.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Other: Sensory Thresold, Burst High Frecuency — The ultrasound guided percutaneous peripheral nerve stimulation will be applied to the Spinal or Inferior Gluteal and Tibial Nerve. The parameters will be 5 trains of 5 seconds, 55 seconds apart, at a frequency of 100Hz, making 5 minutes of total treatment. The intensity will be set 200 microamperes (μA) above the detection threshold for each patient, guaranteeing a sensitive but not painful perception.
  Arms: Sensory Threshold, Burst High Frequency
Other: Theta-Burst Stimulation — The ultrasound guided percutaneous peripheral nerve stimulation will be applied to the Spinal or Inferior Gluteal and Tibial Nerve. The parameters will be 40 trains separated by 7 seconds from each other, where each train contains 5 trains separated by 200ms, at a frequency of 5Hz, resulting in 6 minutes and 45 seconds of total treatment. The intensity will be set at the motor threshold of the patient, ensuring a non-painful stimulation.
  Arms: Theta-Burst Stimulation
Other: Transcutaneous Electrical Nerve Stimulation — The transcutaneous electrical nerve stimulation will be applied on the trapezius or low back and internal calf muscles at a frequency of 80Hz and a pulse width of 250 microseconds, for 15 minutes. The intensity will be set at the detection threshold of each patient generating a sensitive but non-painful perception.
  Arms: Transcutaneous Electrical Nerve Stimulation

SUMMARY:
Percutaneous Peripheral Nerve Stimulation (pPNS) is a physical therapy technique, whose main objective is to treat neuro-musculo-skeletal signs and symptoms by applying a current to a peripheric nerve with a blunt dry needle. Despite its clinical use being already stablished, its use in pathologic subjects is still unknown and, thus, so is its optimal parameterization. The present study proposes to perform two different protocols of peripheral nerve stimulation on neck and low back pain subjects to answer those questions and compared it towards a control group receiving a standard intervention.

DETAILED DESCRIPTION:
Intervention will be performed on the Spinal Nerve (for neck pain subjects) and Inferior Gluteal Nerve and Tibial Nerve (for low back pain subjects), using ultrasonography to guide the needle insertion, without risk of affecting any adjacent structure. The theoretical basis of the technique is to produce analgesia by making controlled changes in the somatosensory system using synaptic plasticity, to ultimate affect the perception of pain through reduction of nociception afference. The protocols will be the following:

* Intervention Group 1: Sensory Threshold, high frequency in trains (ST-bHF). 5 trains of 5 seconds, separated by 55 seconds from each other, at a frequency of 100 hertz (Hz), making 5 minutes of total treatment. The intensity will be set at patient's sensory threshold, ensuring a non-painful perception.
* Intervention Group 2: Theta-Burst Stimulation (TBS). 40 trains separated 10 seconds apart, where each train contains 5 trains separated by 200ms, at a frequency of 5 hertz, resulting in 6 minutes and 45 seconds of total intervention. The intensity will be set at patient's motor threshold, ensuring a non-painful stimulation.
* Intervention Group 3: Transcutaneous electrical nerve stimulation (TENS), at a frequency of 80 hertz and a pulse width of 250 microseconds, for 15 minutes. The intensity will be set at the detection threshold of each patient, generating a sensitive but not painful sensory but not painful.

The study will be a randomised quadruple-blind clinical trial. Two pPNS protocols (ST-bHF, TBS) and a third TENS protocol (TENS) will be compared. To study the effects of these protocols on pain, strength, functionality and electromyographic activity, three measurements will be performed: pre-intervention (Numerical Pain Scale (NRS), NRS for induced pain, Maximal strength + EMG), during the intervention (EMG) and immediately post-intervention (NRS, NRS for induced pain, Maximal strength + EMG). In addition, one week later, subjects will be asked for a pain NRS to assess the mid-term treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Adults (+18 years)
* Patients with non-specific/mechanical/articular neck pain.
* Patients with non-specific/mechanical/articular low back pain and/or low back pain accompanied by radicular symptomatology or sciatica.

Exclusion Criteria:

* Pregnancy.
* Severe illnesses: diabetes, cancer, neurological diseases, depression, etc...
* Balanophora (needle phobia).
* Professional athlete.
* Other concomitant physiotherapy treatment for this pathology.
* Patients with neck or low back pain associated with severe bone damage such as fractures or vertebral fissures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Change in Pain | Pre-intervention and immediately after the intervention
  The subject will verbally report the pain intensity suffered along the last week according to the Numeric rate scale (NRS): 0 will be any pain and 10 will be the maximal perception of pain.

SECONDARY OUTCOMES:
Demographic questionnaire | Pre-intervention
  Patients will fill a demographic data questionnaire with descriptive variables such as age, sex, work, time with pain, concomitant pathologies, level of sporting activity, toxic habits and drugs.
Change in pain | Pre-intervention and one week after the intervention
  The subject will verbally report a mean of the last week pain intensity according to the Numeric rate scale (NRS) from 0 to 10: 0 will be any pain and 10 will be the maximal perception of pain.
  One week after the intervention, and after having received a conventional physiotherapy treatment, subjects will verbally report a mean of the last week pain intensity according to the Numeric rate scale (NRS).
Change in pain evoked with movement | Pre-intervention and immediately after the intervention
  Participants will be asked to perform a motion that evokes pain related to their pathology. After performing the movement, the pain perception will be obtained from 0 to 10 according to the NRS scale: 0 will be any pain and 10 will be the maximal perception of pain.
Change in maximum strength during muscle contraction with dynamometer | Pre-intervention and immediately after the intervention
  The maximum strength achievable given the condition will be assessed by means of a dynamometry test. Neck pain subjects will stand up and perform a maximum voluntary trapezius contraction by raising the shoulder towards the ceiling. Low back pain subjets will be in prone position, resting the trunk on the bed, but no the lower limbs, that will be resting on the floor. They will perform a maximum voluntary unilateral hip extension with the homolateral leg extended and the other leg resting on the floor. In order to not influence the measurement, all subjects will receive the same instructions on how to perform the contraction: "fast and hard", and will be encouraged during the task. Three test will be performed, and a first familiarisation test will be discarded. The rest between measurements will be 1 minute.
Change in surface electromyography signal during muscle contraction | Pre-intervention and immediately after the intervention
  Electrical activity of trapezius muscle (descending fibres) or gluteus maximus muscle will be measured synchronously with strength. Electromyography measurement will be performed in order to collect the muscle excitation signal during the muscle contraction. For the trapezius, electrodes will be placed in the middle of an imaginary line joining prominences of the acromion and C7's spinous apophysis. For the gluteus maximus, the electrodes will be placed in the middle of an imaginary line joining prominences of the sacrum and trochanter.
Surface electromyography signal during stimulation | During intervention
  Electrical activity of trapezius muscle (descending fibres) or gluteus maximus and internal calf muscle will be measured synchronously with treatment application. Electromyography measurement will be performed in order to collect the muscle excitation signal during the electrical stimulation. For the trapezius, the electrodes will be placed in the middle of an imaginary line joining prominences of the acromion and C7's spinous apophysis. For the gluteus maximus, the electrodes will be placed in the middle of an imaginary line joining prominences of the sacrum and trochanter. For the inner calf, a plantar flexion will be requested to the subject to visualize the center of the muscle belly, where the electrodes will be placed.
Treatment-evoked perceptions questionnaire | Immediately after the intervention
  After the stimulation, subjects will be asked about their perceptions related to sensations during stimulation (pleasant- displeasing- indifferent), contraction of the area during the treatment (increasingly- decreasingly- equal), and changes in the strength of the treated area (more- less- equal).

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Velasco Serna, PhD, Principal Investigator — VIB-KULeuven
Locations (1):
- Ionclinics & DEIONICS, Valencia, Spain

REFERENCES:
- [Background] Abejon D, Perez-Cajaraville J. Peripheral nerve stimulation: definition. Prog Neurol Surg. 2011;24:203-209. doi: 10.1159/000323052. Epub 2011 Mar 21. PMID 21422790
- [Background] Bear MF, Malenka RC. Synaptic plasticity: LTP and LTD. Curr Opin Neurobiol. 1994 Jun;4(3):389-99. doi: 10.1016/0959-4388(94)90101-5. PMID 7919934
- [Background] Bevan S. Economic impact of musculoskeletal disorders (MSDs) on work in Europe. Best Pract Res Clin Rheumatol. 2015 Jun;29(3):356-73. doi: 10.1016/j.berh.2015.08.002. Epub 2015 Oct 24. PMID 26612235
- [Background] Borghouts JAJ, Koes BW, Bouter LM. The clinical course and prognostic factors of non-specific neck pain: a systematic review. Pain. 1998 Jul;77(1):1-13. doi: 10.1016/S0304-3959(98)00058-X. PMID 9755013
- [Background] Corp N, Mansell G, Stynes S, Wynne-Jones G, Morso L, Hill JC, van der Windt DA. Evidence-based treatment recommendations for neck and low back pain across Europe: A systematic review of guidelines. Eur J Pain. 2021 Feb;25(2):275-295. doi: 10.1002/ejp.1679. Epub 2020 Nov 12. PMID 33064878
- [Background] Delgado Conforme, W. A., Abarca López, J. J., Boada Rodríguez, L. E., & Salazar Trujillo, S. E. (2019). Lumbalgia inespecífica. Dolencia más común de lo que se cree. RECIMUNDO, 3(2), 3-25. https://doi.org/10.26820/recimundo/3.(2).abril.2019.3-25
- [Background] Ghoname EA, Craig WF, White PF, Ahmed HE, Hamza MA, Henderson BN, Gajraj NM, Huber PJ, Gatchel RJ. Percutaneous electrical nerve stimulation for low back pain: a randomized crossover study. JAMA. 1999 Mar 3;281(9):818-23. doi: 10.1001/jama.281.9.818. PMID 10071003
- [Background] Gutierrez-Muto AM, Castilla J, Freire M, Oliviero A, Tornero J. Theta burst stimulation: Technical aspects about TMS devices. Brain Stimul. 2020 May-Jun;13(3):562-564. doi: 10.1016/j.brs.2020.01.002. Epub 2020 Jan 9. No abstract available. PMID 32289677
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Hjornevik T, Jacobsen LM, Qu H, Bjaalie JG, Gjerstad J, Willoch F. Metabolic plasticity in the supraspinal pain modulating circuitry after noxious stimulus-induced spinal cord LTP. Pain. 2008 Dec;140(3):456-464. doi: 10.1016/j.pain.2008.09.029. Epub 2008 Nov 11. PMID 19004552
- [Background] Huang Y, Chen SR, Chen H, Zhou JJ, Jin D, Pan HL. Theta-Burst Stimulation of Primary Afferents Drives Long-Term Potentiation in the Spinal Cord and Persistent Pain via alpha2delta-1-Bound NMDA Receptors. J Neurosci. 2022 Jan 19;42(3):513-527. doi: 10.1523/JNEUROSCI.1968-21.2021. Epub 2021 Dec 8. PMID 34880118
- [Background] Jauregui JJ, Cherian JJ, Gwam CU, Chughtai M, Mistry JB, Elmallah RK, Harwin SF, Bhave A, Mont MA. A Meta-Analysis of Transcutaneous Electrical Nerve Stimulation for Chronic Low Back Pain. Surg Technol Int. 2016 Apr;28:296-302. PMID 27042787
- [Background] Jimenez S, Mordillo-Mateos L, Dileone M, Campolo M, Carrasco-Lopez C, Moitinho-Ferreira F, Gallego-Izquierdo T, Siebner HR, Valls-Sole J, Aguilar J, Oliviero A. Effects of patterned peripheral nerve stimulation on soleus spinal motor neuron excitability. PLoS One. 2018 Feb 16;13(2):e0192471. doi: 10.1371/journal.pone.0192471. eCollection 2018. PMID 29451889
- [Background] Johnson MI, Paley CA, Jones G, Mulvey MR, Wittkopf PG. Efficacy and safety of transcutaneous electrical nerve stimulation (TENS) for acute and chronic pain in adults: a systematic review and meta-analysis of 381 studies (the meta-TENS study). BMJ Open. 2022 Feb 10;12(2):e051073. doi: 10.1136/bmjopen-2021-051073. PMID 35144946
- [Background] Kazeminasab S, Nejadghaderi SA, Amiri P, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Neck pain: global epidemiology, trends and risk factors. BMC Musculoskelet Disord. 2022 Jan 3;23(1):26. doi: 10.1186/s12891-021-04957-4. PMID 34980079
- [Background] Knezevic NN, Candido KD, Vlaeyen JWS, Van Zundert J, Cohen SP. Low back pain. Lancet. 2021 Jul 3;398(10294):78-92. doi: 10.1016/S0140-6736(21)00733-9. Epub 2021 Jun 8. PMID 34115979
- [Background] Lall MP, Restrepo E. The Biopsychosocial Model of Low Back Pain and Patient-Centered Outcomes Following Lumbar Fusion. Orthop Nurs. 2017 May/Jun;36(3):213-221. doi: 10.1097/NOR.0000000000000350. PMID 28538537
- [Background] Larson J, Munkacsy E. Theta-burst LTP. Brain Res. 2015 Sep 24;1621:38-50. doi: 10.1016/j.brainres.2014.10.034. Epub 2014 Oct 27. PMID 25452022
- [Background] Larson J, Wong D, Lynch G. Patterned stimulation at the theta frequency is optimal for the induction of hippocampal long-term potentiation. Brain Res. 1986 Mar 19;368(2):347-50. doi: 10.1016/0006-8993(86)90579-2. PMID 3697730
- [Background] Lin T, Gargya A, Singh H, Sivanesan E, Gulati A. Mechanism of Peripheral Nerve Stimulation in Chronic Pain. Pain Med. 2020 Aug 1;21(Suppl 1):S6-S12. doi: 10.1093/pm/pnaa164. PMID 32804230
- [Background] Luo C, Kuner T, Kuner R. Synaptic plasticity in pathological pain. Trends Neurosci. 2014 Jun;37(6):343-55. doi: 10.1016/j.tins.2014.04.002. Epub 2014 May 12. PMID 24833289
- [Background] Maffiuletti NA, Aagaard P, Blazevich AJ, Folland J, Tillin N, Duchateau J. Rate of force development: physiological and methodological considerations. Eur J Appl Physiol. 2016 Jun;116(6):1091-116. doi: 10.1007/s00421-016-3346-6. Epub 2016 Mar 3. PMID 26941023
- [Background] Martimbianco ALC, Porfirio GJ, Pacheco RL, Torloni MR, Riera R. Transcutaneous electrical nerve stimulation (TENS) for chronic neck pain. Cochrane Database Syst Rev. 2019 Dec 12;12(12):CD011927. doi: 10.1002/14651858.CD011927.pub2. PMID 31830313
- [Background] Plaza-Manzano G, Gomez-Chiguano GF, Cleland JA, Arias-Buria JL, Fernandez-de-Las-Penas C, Navarro-Santana MJ. Effectiveness of percutaneous electrical nerve stimulation for musculoskeletal pain: A systematic review and meta-analysis. Eur J Pain. 2020 Jul;24(6):1023-1044. doi: 10.1002/ejp.1559. Epub 2020 Apr 4. PMID 32171035
- [Background] Popescu A, Lee H. Neck Pain and Lower Back Pain. Med Clin North Am. 2020 Mar;104(2):279-292. doi: 10.1016/j.mcna.2019.11.003. Epub 2019 Dec 20. PMID 32035569
- [Background] Rampazo EP, Martignago CCS, de Noronha M, Liebano RE. Transcutaneous electrical stimulation in neck pain: A systematic review and meta-analysis. Eur J Pain. 2022 Jan;26(1):18-42. doi: 10.1002/ejp.1845. Epub 2021 Aug 3. PMID 34288255
- [Background] Ranck JB Jr. Studies on single neurons in dorsal hippocampal formation and septum in unrestrained rats. I. Behavioral correlates and firing repertoires. Exp Neurol. 1973 Nov;41(2):461-531. doi: 10.1016/0014-4886(73)90290-2. No abstract available. PMID 4355646
- [Background] Rudell AP, Fox SE, Ranck JB Jr. Hippocampal excitability phase-locked to the theta rhythm in walking rats. Exp Neurol. 1980 Apr;68(1):87-96. doi: 10.1016/0014-4886(80)90068-0. No abstract available. PMID 7363990
- [Background] Svendsen F, Tjolsen A, Hole K. LTP of spinal A beta and C-fibre evoked responses after electrical sciatic nerve stimulation. Neuroreport. 1997 Nov 10;8(16):3427-30. doi: 10.1097/00001756-199711100-00002. PMID 9427300
- [Background] Van Breukelen GJ. ANCOVA versus change from baseline: more power in randomized studies, more bias in nonrandomized studies [corrected]. J Clin Epidemiol. 2006 Sep;59(9):920-5. doi: 10.1016/j.jclinepi.2006.02.007. Epub 2006 Jun 23. PMID 16895814
- [Background] Wall PD, Sweet WH. Temporary abolition of pain in man. Science. 1967 Jan 6;155(3758):108-9. doi: 10.1126/science.155.3758.108. PMID 6015561
- [Background] Wu J, Hu Q, Huang D, Chen X, Chen J. Effect of electrical stimulation of sciatic nerve on synaptic plasticity of spinal dorsal horn and spinal c-fos expression in neonatal, juvenile and adult rats. Brain Res. 2012 Apr 11;1448:11-9. doi: 10.1016/j.brainres.2012.02.002. Epub 2012 Feb 13. PMID 22377455
- [Background] Yang F, Guo J, Sun WL, Liu FY, Cai J, Xing GG, Wan Y. The induction of long-term potentiation in spinal dorsal horn after peripheral nociceptive stimulation and contribution of spinal TRPV1 in rats. Neuroscience. 2014 Jun 6;269:59-66. doi: 10.1016/j.neuroscience.2014.03.037. Epub 2014 Mar 26. PMID 24680883
- [Derived] Ortega FJ, Giner MJ, Perez-Cervera L, Tomas E, Valdesuso R, Navarro I, Delicado-Miralles M, Velasco E. Plasticity-Inducing Percutaneous Peripheral Nerve Stimulation for Treating Neck Pain: A Blinded, Randomised Clinical Trial. Eur J Pain. 2026 Jan;30(1):e70207. doi: 10.1002/ejp.70207. PMID 41555668